CLINICAL TRIAL: NCT01493986
Title: Minimum Effective Volume of Ropivacaine 7.5 mg/ml for the Lateral and Sagittal Infraclavicular Brachial Plexus Block When Using Guidance by Both Ultrasound and Nerve Stimulation.
Brief Title: Minimum Effective Volume of Ropivacaine 7.5 mg/ml for the Lateral and Sagittal Infraclavicular Brachial Plexus Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Lars Marius Ytrebo, Professor, University Hospital of North Norway
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UNorthNorway
Record Dates: First submitted 2011-12-14; First posted 2011-12-16 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Pain
Keywords: Ropivacaine; Brachial plexus
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ropivacaine — Dosage. Onset time
  Other Names: Naropin

SUMMARY:
Systemic LA toxicity is an important complication of regional anesthesia. Lowering the LA dose is one of the strategies to reduce this risk. For upper limb blocks it is well documented that ultrasound guidance allows a significant lower dose of LA for interscalene and axillary blocks than with guidance by peripheral nerve stimulation. However, a corresponding difference has not yet been found for supraclavicular and infraclavicular blocks. The aim of the present study is to define the minimum effective volume of ropivacaine 7.5 mg/ml when using the LSIB method.

DETAILED DESCRIPTION:
The blocks will be performed as previously described, by an anesthesiologist with LSIB expertise. The lateral, medial and posterior cords are the target of infra-clavicular brachial plexus blocks. During a prescan we will record if they can be visualized by ultrasound and indicate their positions periarterially. The deep location of the cords may hamper their identification, especially that of the medial cord. We describe the cord positions with reference to the short-axis (cross-sectional) view of the axillary artery, which is compared to a clockface having 12 o'clock ventrally. In a former MRI study it was found that the cords were usually located in a sector from 3-11 o'clock (the 3-11 sector) and within a distance of 2 cm from the midaxis of the axillary artery. The point closest to the cords was at 8 o'clock, immediately outside the arterial wall. Point of needle insertion is at the intersection between the lower edge of the clavicle and the medial surface of the coracoid process. We direct the needle tip to the 8 o'clock position and observe the spread of LA from this position. On demand we adjust the needle position to secure a complete fill of the 3-11 sector with LA (multiple injections).

The block needle has an electrical cable. Prior to LA injections we test if a minimal electric output (0.2 mA/0.1 msec duration) elicits a motor response. If such a response is obtained, the needle is withdrawn (in steps of 1 mm), until the motor response disappears. This is to reduce the risk of intraneural injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients of American Society of Anesthesiologists physical status (ASA) I-II
* Scheduled for surgery distal to the elbow.
* Duration of surgery >1 hour.
* Age 18-65 years,
* Body mass index 20-35 kg/m2

Exclusion Criteria:

* Pregnancy
* Any contraindication to regional anesthesia
* Patients on major opioids because of chronic pain
* Atrioventricular block
* Pacemaker
* Diabetes
* Peripheral neuropathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the minimum effective volume of ropivacaine 7.5 mg/ml providing a successful infraclavicular block (LSIB) in 50% of the patients (MEAV50). | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Lars M Ytrebo, Professor, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway